CLINICAL TRIAL: NCT04457778
Title: Phase I, First-in-Human, Open-Label, Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Clinical Activity of M6223, an Inhibitor of TIGIT, as Single Agent and in Combination With Bintrafusp Alfa (Anti-PDL1/ TGFß Trap) in Participants With Metastatic or Locally Advanced Solid Unresectable Tumors
Brief Title: First in Human Study of M6223
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS201430_0001
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Solid Tumors
Keywords: M6223; Bintrafusp alfa; Metastatic Solid Tumors
MeSH Terms: interventions — bintrafusp alfa protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1A: M6223 Monotherapy (Experimental)
  Interventions: Drug: M6223
- Part1B: M6223 + Bintrafusp alfa (Experimental)
  Interventions: Drug: Bintrafusp alfa; Drug: M6223

INTERVENTIONS:
Drug: M6223 — Participants will receive an intravenous (IV) infusion of M6223 at escalated doses every 2 weeks (Q2W) or every 3 weeks (Q3W) on Day 1 of each Cycle (Each cycle is of 14 days) according to the recommendation of the SMC(Safety Monitoring Committee) until the maximum tolerated dose(MTD) has been reached or confirmed disease progression.
  Arms: Part 1A: M6223 Monotherapy
Drug: Bintrafusp alfa — Participants will receive an IV infusion of bintrafusp alfa Q2W on Day 1 of each Cycle (Cycle is 14 days) until confirmed disease progression.
  Arms: Part1B: M6223 + Bintrafusp alfa
Drug: M6223 — Participants will receive an IV infusion of M6223 at escalated doses Q2W on Day 1 of each Cycle (Each cycle is of 21 days) according to the recommendation of the SMC until the MTD has been reached or confirmed disease progression.
  Arms: Part1B: M6223 + Bintrafusp alfa

SUMMARY:
The main purpose of this study is to determine the safety, tolerability, pharmacokinetics (PK), immunogenicity and (if observed) the maximum tolerated dose (MTD) of M6223 as a single agent (Part 1A) for both the every 2 weeks (Q2W) regimen and the every 3 weeks (Q3W) regimen and of M6223 combined with bintrafusp alfa (Part 1B) for Q2W regimen in participants with metastatic or locally advanced solid unresectable tumors.

ELIGIBILITY:
Inclusion Criteria:

* Participants have histologically or cytologically proven locally advanced or advanced solid malignancies who are refractory to or have progressed under standard treatment and have no other treatment options known to confer clinical benefit
* Participants with Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 1 at Screening
* Participant has a formalin-fixed paraffin-embedded block containing tumor tissue or a minimum of 15 (preferably 25) unstained tumor slides suitable for immunohistochemistry-based staining of protein expression
* Participants with life expectancy of at least 12 weeks
* Participants with measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)
* Adequate hematological, hepatic and renal function as defined in the protocol
* Other protocol defined inclusion criteria may apply

Exclusion Criteria:

* Participants with persisting toxicity related to prior therapy Grade greater than (>) 1 National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0, however, alopecia, sensory neuropathy Grade less than or equal to (<=) 2, or other non-immune-related Grade <= 2 not constituting a safety risk
* Participants with prior organ transplantation including allogeneic stem cell transplantation
* Participants with prior toxicity related to an immune checkpoint inhibitor Grade greater than equal to (>=) 3 NCI-CTCAE Version 5.0 unless resolved to Grade <= 1 prior to study inclusion
* Participants with current significant cardiac conduction abnormalities, including corrected QT interval (QTcF, corrected with Fridericia formula) prolongation of > 450 milli seconds (ms) on triplicate 12-lead ECG or impaired cardiovascular function, ventricular tachycardia, hypokalemia or a history of paroxysmal atrial fibrillation, serious cardiac arrhythmia and family history of sudden death or long QT syndrome
* A history of vascular, cardiovascular or cerebrovascular disease like, cerebral vascular accident/stroke (less than [<] 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class >= II), deep vein thrombosis (< 3 months prior to enrollment) or pulmonary thrombosis/embolism (< 3 months prior to enrollment)
* Other protocol defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-06-23 (Actual)

PRIMARY OUTCOMES:
Part 1A and 1B: Occurrence of Dose Limiting Toxicities (DLTs) During the DLT Observation Period (28 Days) | Day 1 to Day 28
Part IA and IB: Occurrence of Treatment-Emergent Adverse Events (TEAEs) and Treatment Related Adverse Events (TRAEs) According to the National Cancer Institute Common Terminology Criteria of Adverse Events (NCI-CTCAE) version 5 | Time from first study drug administration to final assessment at end of safety follow-up visit (up to a maximum of approximately 2 years)
Part IA and IB: Occurrence of Treatment-Emergent Adverse Events (TEAEs) as per Severity and Deaths | Time from first study drug administration to final assessment at end of safety follow-up visit (up to a maximum of approximately 2 years)
Part IA and IB: Occurrence of Clinically Significant Change From Baseline in Clinical Laboratory Measures | Time from baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 2 years)
Part IA and IB: Occurrence of Clinically Significant Change From Baseline in Electrocardiogram Findings | Time from baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 2 years)
Part IA and IB: Occurrence of Clinically Significant Change From Baseline in Vital Signs | Time from baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 2 years)
Part IA and IB: Occurrence of Change From Baseline in Eastern Cooperative Oncology Group Performance Status | Time from baseline to final assessment at end of safety follow-up visit (up to a maximum of approximately 2 years)

SECONDARY OUTCOMES:
Part 1A and Part 1B: Area Under the Serum Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC 0-t) of M6223 | Pre-dose up to 14 days (in Q2W regimen) or 21 days (in Q3W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen and each Cycle is of 21 days in Q3W regimen)
Part 1A and Part 1B: Area Under the Serum Concentration-Time Curve From Time Zero to Infinity (AUC 0-inf) of M6223 | Pre-dose up to 14 days (in Q2W regimen) or 21 days (in Q3W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen and each Cycle is of 21 days in Q3W regimen)
Part 1A and Part 1B: Area Under Serum Concentration-Time Curve Over a Dosing Interval From Time Zero to Tau (τ) (AUCτ) of M6223 | Pre-dose up to 14 days (in Q2W regimen) or 21 days (in Q3W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen and each Cycle is of 21 days in Q3W regimen)
Part 1A and Part 1B: Maximum Observed Serum Concentration (Cmax) of M6223 | Pre-dose up to 14 days (in Q2W regimen) or 21 days (in Q3W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen and each Cycle is of 21 days in Q3W regimen)
Part 1A and Part 1B: Serum Concentration Observed Immediately Before Next Dosing (Ctrough) of M6223 | Pre-dose up to 14 days (in Q2W regimen) or 21 days (in Q3W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen and each Cycle is of 21 days in Q3W regimen)
Part 1A and Part 1B: Time to Reach Maximum Serum Concentration (Tmax) of M6223 | Pre-dose up to 14 days (in Q2W regimen) or 21 days (in Q3W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen and each Cycle is of 21 days in Q3W regimen)
Part 1A and Part 1B: Apparent Terminal Half-Life (t1/2) of M6223 | Pre-dose up to 14 days (in Q2W regimen) or 21 days (in Q3W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen and each Cycle is of 21 days in Q3W regimen)
Part 1A and Part 1B: Elimination Rate Constant (Lambda z) of M6223 | Pre-dose up to 14 days (in Q2W regimen) or 21 days (in Q3W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen and each Cycle is of 21 days in Q3W regimen)
Part 1B: Maximum Observed Serum Concentration (Cmax) of Bintrafusp alfa | Pre-dose up to 14 days (in Q2W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen)
Part 1B: Serum Concentration Observed Immediately Before Next Dosing (Ctrough) of Bintrafusp alfa | Pre-dose up to 14 days (in Q2W regimen) post-dose of Cycles 1, 2, and 4 (Each cycle is of 14 days in Q2W regimen)
Part IA and 1B: Immunogenicity of M6223 Measured by Antidrug Antibody (ADA) Assays | Pre-dose of Day 1 Cycle 1 (Each Cycle is of 14 days in Q2W regimen and 21 days in Q3W regimen) up to end of safety follow-up visit (up to a maximum of 2 years)
Part 1B: Immunogenicity of Bintrafusp alfa Measured by Antidrug Antibody (ADA) Assays | Pre-dose of Day 1 Cycle 1 (Each Cycle is of 14 days in Q2W regimen) up to end of safety follow-up visit (up to a maximum of 2 years)
Part 1A and 1B: Change from Baseline in QT Interval | From Day 1 Cycle 1 (Baseline) up to Day 1 Cycle 7 (Each Cycle is of 14 days in Q2W regimen and 21 days in Q3W regimen)
Part 1A and IB: Best Overall Response According to Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed as per Investigator | From first study drug administration until documented disease progression or death due to any cause whichever occurs first, (approximately assessed up to 2 years)
Part 1A and 1B: Duration of Response According to Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed as per Investigator | From first study drug administration until documented disease progression or death due to any cause whichever occurs first, (approximately assessed up to 2 years)
Part 1A and 1B: Time to Tumor Response According to Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed as per Investigator | From first study drug administration until documented disease progression or death due to any cause whichever occurs first, (approximately assessed up to 2 years)
Part 1A and 1B: Disease Control According to Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed as per Investigator | From first study drug administration until documented disease progression or death due to any cause whichever occurs first, (approximately assessed up to 2 years)
Part 1A and 1B: Progression-free Survival Time According to Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Assessed as per Investigator | From first study drug administration until documented disease progression or death due to any cause whichever occurs first, (approximately assessed up to 2 years)
Part 1A and 1B: Overall Survival | Time from first treatment to end of study (planned 12 months after last patient started treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (4):
- United States (3):
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- [Derived] Naing A, McKean M, Tolcher A, Victor A, Hu P, Gao W, Nogueira Filho MAF, Kitzing T, Gleicher S, Holland D, Richter E, Tadjalli-Mehr K, Siu LL. TIGIT inhibitor M6223 as monotherapy or in combination with bintrafusp alfa in patients with advanced solid tumors: a first-in-human, phase 1, dose-escalation trial. J Immunother Cancer. 2025 Feb 10;13(2):e010584. doi: 10.1136/jitc-2024-010584. PMID 39929671
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201430_0001
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: INTR@PID Clinical Trial Program — https://www.intrapidclinicaltrials.com/en